CLINICAL TRIAL: NCT06238323
Title: Adaptation and Feasibility of Many Men Many Voices (3MV), an HIV Prevention Intervention to Reduce Intersectional Stigma and Increase HIVST Among YSMM Residing in Ghanaian Slums - A Clustered Pre-post Pilot Trial Protocol
Brief Title: Lafiya HIV Self-testing Study Protocol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: University of Ghana (Other); George Washington University (Other); Yale University (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Gamji Rabiu Abu-Ba'are, Assistant professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00008385; R01TW012671 (NIH)
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: HIV Prevention and Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): Participants will be young sexual minority men (YSMM) and providers from healthcare institutions working with YSMM.
  Interventions: Behavioral: LAFIYA

INTERVENTIONS:
Behavioral: LAFIYA — LAFIYA will be a modified version of the Many Men Many Voices (3MV) targeted at addressing reducing stigma and increasing HIV self-testing uptake among young sexual minority men. LAFIYA will be developed into a comprehensive intervention manual for a large-scale trial using the ADAPTT-IT framework.

SUMMARY:
The study aims to address low testing and related issues such as stigma, low-risk perception, and concerns about confidentiality affecting testing. To overcome these challenges, the study proposes to adapt the Many Men Many Voices (3MV) into a modified version called LAFIYA to tackle intersectional stigma and improve HIVST among young sexual minority men in Ghana.

ELIGIBILITY:
Inclusion Criteria:

* YSMM: To be eligible to participate in the interview, the person must be between 18 to 25 years old, have no experience using unassisted HIVST kits, do not know their HIV status or tested negative, currently identifies as cis-gender man, and have had sex with another man within six months before engaging with the recruitment team and must reside within a slum community in the Greater Accra Metropolitan area.
* Providers: To be eligible to participate in the interview, the person must have experience providing sexual health services such as HIV testing, counseling, and linkage to prevention and care services for at least one year. Must reside within the Greater Accra Metropolitan area and have worked with YSMM on HIV prevention and care.

Exclusion Criteria:

* YSMM: Those who fall under 18 years or above 25 years will be excluded from the study. YSMM who have experience with unassisted HIVST kits, know their HIV status, or tested positive for HIV will be excluded from the study. YSMM who do not identify as cis-gender man and have not had sex with another man within six months before engaging with the recruitment team will be excluded from the study. YSMM who do not reside within a slum community in the Greater Accra Metropolitan area will be excluded from the study.
* Providers: Persons who do not have experience providing services such as HIV testing, counseling, and linkage to prevention and care services for at least one year will be excluded from the study. Providers not residing within the Greater Accra Metropolitan area and have not worked with YSMM on HIV prevention and care will be excluded.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in percentage of participants that reported the intervention as acceptable | Baseline to 3 months
  Participants will be provided with a survey that inquires if HIVST meets their approval, meets their needs, and if they welcome the use of HIVST. Participants will answer yes or no, and reported is the change in the percentage of participants that answered yes to each question.
Change in percentage of participants that reported the intervention as appropriate | Baseline to 3 months
  Participants will be provided with a survey that inquires if HIVST seems reasonable, if HIVST seems like a good match, and if HIVST seems applicable. Participants will answer yes or no, and reported is the change in the percentage of participants that answered yes to each question.
Change in percentage of participants that reported the intervention as feasible. | Baseline to 3 months
  Participants will be provided with a survey that inquires if HIVST seems easy to use, if HIVST seems challenging, and if HIVST seems practical. Participants will answer yes or no, and reported is the change in the percentage of participants that answered yes to each question.

SECONDARY OUTCOMES:
Change in the number of HIV tests | Baseline to 3 months
  We are going to collect the total number of HIV tests performed by all participants and report the mean change in number.
Mean change in the Basic Needs Satisfaction Scale. | Baseline to 3 months
  The Basic Needs Satisfaction scale is a 9 question scale that asks participants general questions about experiences of feeling free within their community while identifying as YSMM. The outcome measure will analyze changes in average scores over time. The Basic Needs Satisfaction Scale is scored on a scale ranging from 1 to 10, where 1 represents the lowest possible level of basic needs satisfaction, and 10 represents the highest
Percentage of participants to report resilience/bouncing back after hard times. | Baseline to 3 months
  Participants will be provided with a 6 question survey that inquires into a percentage change in their level of resilience. Each question inquires into their ability to bounce back or cope with challenges, with responses categorized as "yes" or "no." The survey results are then analyzed by calculating the percentage of participants who responded affirmatively (yes) to each question. The average percentage across all questions is calculated to arrive at an overall percent score.
Percentage of participants that reported enacted stigma. | Baseline to 3 months
  Participants will be provided with a 10 question survey that inquires into the rate at which they experienced unfair treatment by others. Each question will inquire into experiences of unfair treatment, with responses categorized as "yes" or "no." The survey results are then analyzed by calculating the percentage of participants who responded affirmatively (yes) to each question. The average percentage across all questions is calculated for an overall percent score.
Percentage of participants that reported vicarious stigma. | Baseline to 3 months
  Participants will be provided with a 10 question survey that inquires into the percentage rate at which they have heard stories about other YSMM stigma experiences. Each question inquires whether they have heard stories of other YSMM experiencing stigma, with responses categorized as "yes" or "no." The survey results are then analyzed by calculating the percentage of participants who responded affirmatively (yes) to each question. The average percentage across all questions is calculated to arrive at an overall percent score.
Percentage of participants that reported perceived stigma. | Baseline to 3 months
  Participants will be provided with a 10 question survey that inquires into the level of agreement or disagreement on perceived stigma. Each question inquires whether they agree or disagree with perceived stigma, with responses categorized as "yes" or "no." The survey results are then analyzed by calculating the percentage of participants who responded affirmatively (yes) to each question. The average percentage across all questions is calculated to arrive at an overall percent score.
Percentage in participants that reported internalized stigma. | Baseline to 3 months
  Participants will be provided with a 10 question survey that inquires into the percentage change in internalized stigma. Each question inquires into their experience of internalized stigma, with responses categorized as "yes" or "no." The survey results are then analyzed by calculating the percentage of participants who responded affirmatively (yes) to each question. The average percentage across all questions is calculated to arrive at an overall percent score.
Percentage of participants that reported stigma for involving in same sex relations. | Baseline to 3 months
  Participants will be provided with a 10 question survey that inquires into the frequency at which they encounter stigma from engaging in same-sex relations. Each question inquires into their experiences of stigma from engaging in same-sex relationships, with responses categorized as "yes" or "no." The survey results are then analyzed by calculating the percentage of participants who responded affirmatively (yes) to each question. The average percentage across all questions is calculated to arrive at an overall percent score.
Percentage of participants that reported stigma from being gender non-conforming. | Baseline to 3 months
  Participants will be provided with a 10 question survey that inquires into the frequency at which they encounter stigma due to their feminine mannerisms. Each question inquires into their experiences of stigma from being gender non-conforming, with responses categorized as "yes" or "no." The survey results are then analyzed by calculating the percentage of participants who responded affirmatively (yes) to each question. The average percentage across all questions is calculated to arrive at an overall percent score.
Healthcare climate | Baseline to 3 months
  Participants will be provided with a 6 question survey that inquires into the frequency at which they encounter negative health provider attitudes. Each question inquires into their experiences when dealing with health providers, with responses categorized as "yes" or "no." The survey results are then analyzed by calculating the percentage of participants who responded affirmatively (yes) to each question. The average percentage across all questions is calculated to arrive at an overall percent score.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ghana, Accra, Ghana

IPD SHARING:
Plan to Share IPD: No